CLINICAL TRIAL: NCT06560437
Title: Effects of the Chinese Jingjin Manual Therapy on Brain Function in Young Cervical Spondylosis Patients With Chronic Neck Pain: an fMRI Study
Brief Title: Effects of the Manual Therapy on Brain Function in Young Chronic Neck Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wendi Zhang (Other)
Responsible Party: Sponsor-Investigator, Wendi Zhang, Chinese Medicine Sinew Injury Clinic Doctor, The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Organization: The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023AH-17
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the CNP group (Experimental): The CNP group received Chinese Jingjin manual therapy which is divided into three major parts: fascia manipulation, bone setting manipulation, and finishing techniques. The operation takes about 30 minutes, and there is one treatment every other day, three treatments per week, and five consecutive weeks of treatment.
  Interventions: Other: Chinese Jingjin Manual Therapy
- the HC groups (No Intervention): The healthy control group without intervention

INTERVENTIONS:
Other: Chinese Jingjin Manual Therapy — Chinese Jingjin therapy is a form of manual therapy that utilizes the principles of Chinese Jingjin Theory (also known as Chinese Sinew Channel Theory) to alleviate nodular lesions in sinew channels caused by Jingjin injuries and to realign skeletal joints. Chinese Jingjin manual therapy is divided into three major parts: fascia manipulation, bone setting manipulation, and finishing techniques. The operation takes about 30 minutes, and there is one treatment every other day, three treatments per week, and five consecutive weeks of treatment.
  Other Names: Chinese Sinew Manual Therapy
  Arms: the CNP group

SUMMARY:
The goal of this clinical trial is to study the central remodeling mechanism of young chronic neck pain patients based on resting-state functional magnetic resonance, and also to study the central analgesic mechanism of Chinese Jingjin Manual Therapy in treating young chronic neck pain patients. The main question it aims to answer are:

Are there specific differences in functional brain activities between young chronic neck pain patients and healthy volunteers? Are there specific changes in brain network function in young chronic neck pain patients before and after Chinese Jingjin Manual Therapy?

Participants will:

The patients in the neck pain group will receive Chinese Jingjin Manual Therapy three times a week for five consecutive weeks.

Before and after the Chinese Jingjin Manual Therapy, patients in the neck pain group were assessed by pressure pain threshold, Northwick Park Questionnaire, and Hospital Anxiety and Depression Scale.

In addition, resting-state functional magnetic resonance data will be collected from the neck pain group and the healthy control group.

DETAILED DESCRIPTION:
Chronic neck pain (CNP) is a prevalent condition of the musculoskeletal system that seriously impacts patients' quality of life. The safety and efficacy of Chinese Jingjin manual therapy, a characteristic of Chinese medicine rehabilitation therapy, have been widely recognized. Its mechanism of action is believed to be associated with the functional modulation of brain region networks.Based on the resting-state functional magnetic resonance imaging (fMRI) amplitude of low-frequency fluctuation (ALFF) technique, to observe the differences in spontaneous activity of brain regions between young CNP patients and healthy people. Additionally, the study aims to investigate the changes in brain network function prior to and following the administration of Chinese Jingjin manual therapy.

ELIGIBILITY:
Inclusion Criteria:

Compliance with the diagnostic basis of cervical spondylosis in the Expert Consensus on Typology, Diagnosis, and Nonsurgical Treatment of Cervical Spondylosis issued by China in 2018 and the Diagnostic Efficacy Criteria for Chinese Medicine issued by State Administration of Traditional Chinese Medicine in 2018.

Neck pain is the main symptom lasting over 12 weeks. Between the ages of 18 and 44 and be right-handed. Had not received treatment for neck pain within the past month. Voluntary participation in the study, ability to complete the entire treatment program, and signing the informed consent form.

Exclusion Criteria:

The condition was in the acute phase stage (within two weeks of onset). Neck pain is caused by other diseases such as fracture, dislocation, and infection.

Severe heart, liver, kidney, and other vital organ diseases or cognitive impairment.

Pregnant or lactating women, severe osteoporosis. Metal foreign bodies in the body or other contraindications to fMRI examination.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Amplitude of low-frequency fluctuation value | 5 weeks
  The amplitude of low-frequency fluctuation as a measure of the intensity of spontaneous activity in resting brain regions.
Tenderness threshold | 5 weeks
  The tenderness threshold a test of the maximum pain threshold that the patient can tolerate
Northwick Park Questionnaire | 5 weeks
  The NPQ is a commonly used scale to assess functional impairment in patients with CNP. The lowest score is 0 and the highest score is 36. Higher scores indicate more severe neck dysfunction in the patient.
Hospital Anxiety and Depression Scale | 5 weeks
  The HADS scale can simultaneously assess the anxiety and depression status of CNP patients. The lowest score is 0 and the highest score is 52. The higher the score, the more severe the patient's emotional problems of anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Wendi Zhang, Principal Investigator — Anhui University of Chinese Medicine
Locations (1):
- Wendi Zhang, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes
There are plans to make individual participant data collected in this study such as study protocols and study reports available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: Review request information may be submitted to the principal investigator if researching content in similar fields will be shared.